CLINICAL TRIAL: NCT02410291
Title: Empowering Patients Through Education- Online, Written, and Personal Education Resource for Prostate Cancer Patients Who Need Radiation Therapy to Ensure Patient Preparedness (Compliance and Understanding) for Their Simulation and Treatment
Brief Title: Impact on Instructional Video on Patients' Compliance With Preparation During CT Planning for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Krista Dawdy, Clinical Educator, Radiation Therapy, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sunnybrook ID 123
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Latent Cancer (Prostate)

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients will receive the standard are to prepare them for their planning CT scan. They will be presented with the flyer that will be developed based on information about the importance of rectal and bladder preparation that is currently provided to patients and will also watch a youtube video on how to prepare for their CT simulation appointment. A few days before the CT planning appointment, patients in this group will be called by the radiation therapist or RA, reminding them about the rectal preparation for the appointment. Each patient will also be reminded to watch the instructional video on YouTube. Patients will be asked not to share the video link with other patients during the study.
  Interventions: Other: Educational video
- Control group (No Intervention): Patients in this group will receive the standard care to prepare them for their planning CT scan. They will be presented with the flyer at the consultation. A few days before the CT appointment, patients in this group will also be called and reminded about the required preparations, but will not be told about the video. In addition to the statistics about patient preparedness collected by the radiation therapist conducting the CT scan and stored and secured in an OCC Pinnacle planning system, we will also evaluate: patients' satisfaction with the preparation instructions, their knowledge (knowledge questionnaire) about the video content and importance of understanding the rectal emptying procedures, and radiation therapists' satisfaction with patients' rectal preparation.

INTERVENTIONS:
Other: Educational video — Patients in the control group will receive standard patient education Patients in the experimental group will receive standard education and an educational video
  Arms: Experimental group

SUMMARY:
Rectal toxicity limits dose escalated intensity modulated radiotherapy (IMRT) for prostate cancer. The dose volume constraints that predict for rectal toxicity require minimizing prostate motion and rectum and bladder filling of IMRT .5-15 . The volumetric changes and internal organ motion during prostate IMRT increases risk of PSA failure in patients with large rectums at the planning CT scans. Patient preparation for IMRT planning is crucial .The literature is limited regarding the effectiveness of educational intervention with behavioral reinforcement for patients, and a gap if exists literacy level is considered. Patients often cannot comprehend verbal or written instructions and have difficulties following through with recommended regimens.23 Using multimedia such as Internet, audio-visual media such as DVD and even the telephone can enhance patients' knowledge and understanding about importance of preparation for IMRT for prostate ca. Thomas's study showed that in patients undergoing radiotherapy and chemotherapy, the video group had lower anxiety scores compared with the non video group. At SOCC patients have been provided with verbal information about bladder and rectum preparation for prostate planning CT scan and IMRT. Patients should have a "fullish" bladder and empty rectum at the time of CT simulation. If the rectal diameter is > 4cm, the patient will be asked to empty his stool/gas and re-scanned. The 3- months review of patients preparedness for prostate IMRT showed that only 13/55 patients were adequately prepared but 42/55 (76%) of patients needed to be re-scanned due to inadequate bladder (21/42, 50%) or rectum filling 28/42, 67%) . Also, 2/13 (15%) patients were still not prepared at the second resimulation despite that they received a phone call with the instructions. The investigators plan to investigate if a multimedia education strategy will decrease costly resimulation rate for patients with prostate cancer.

DETAILED DESCRIPTION:
An estimated 23,600 men will be diagnosed with prostate cancer in Canada in 2014. This represents 24% of all new cancer cases in men in 2014. The SOCC treats 1000 patients with prostate cancer annually. Patients who fail to follow instructions for the initial prostate planning CT scan need to return to be rescanned at a later date. Additional CTs can increase patients' parking and transportation costs and may increase their anxiety. Rescanning may also cause stress to radiation therapists due to unsuccessful planning, increase costs to the cancer centre for the additional time of radiation therapists and increase the planning CT wait time for other patients. Thus improving patients' preparedness for the prostate planning CT scan will reduce costs for patients and the hospital, reduce anxiety and stress for both patients and practitioners, reduce CT scan wait times, maximize the accuracy of prostate IMRT. In a study of 220 patients receiving chemotherapy or radiotherapy, Thomas used video education and the Hospital Anxiety and Depression Scale (HAD) and found a significant correlation between satisfaction and reduced overall treatment related anxiety in the video group22.

Purpose To determine the effectiveness of the introduction of a video on patient preparedness for patients receiving a CT Scan for radiotherapy to the prostate.

Methods The project will consist of three phases: video production, experiment and data collection, and analysis and dissemination.

1. Video production - The investigators will produce the instructional video, test the video, and revise based on initial feedback. Christopher Townsend and Sunnybrook Media will produce the video using the script written by Agnes Ryzynski, with input from team members. The script will highlight the importance of rectal and bladder preparation prior and during the planning CT scans. Images will be presented showing both normal and abnormal preparation examples, instructing patients how to prepare for the planning CT scan. The video will be tested by patients and radiation oncologists, nurses and radiation therapists prior to launch.
2. Experiment and data collection - The investigators will use a control experimental group design. The RA will recruit sixty participants at their pre-planning appointment date or via telephone. The RA will present the study rationale; those who agree to participate will sign the study consent, and be assigned a study entry number. Participants will be randomly assigned to either the control group or the experimental group. The sample size was calculated based on the observed proportion of patients needed to be rescanned: 0.76 (42/55). To have a treatment group with a proportion of 0.38 who needed to be rescanned, a 50% decrease, the investigators will need at least 25 patients in each group to have a power of 0.8, given a 0.05 significance level. To account for study attrition (no more than 20% loss of participants), the investigators will require 30 subjects per group to observe a large treatment effect (e.g. 50% decreases in the proportion of rescanning).
3. Data analysis and dissemination - A statistical analysis will be conducted on the patient preparedness data. The investigators will conduct quantitative analysis of the evaluations form using a Likert scale. Patients' evaluations will also contain open ended questions to capture patients' comments about their experiences during the study. The investigators will analyze the details about patients' and radiation therapists' satisfaction and patients' knowledge about the video content.

Confidentiality Patient confidentiality will be assured. All patients will have assigned a study number and their names will not be disclosed at any time. All study data will be kept in a locked cabinet, that only the investigators have access to.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. All patients who are referred for planning simulation for prostate cancer IMRT will be invited to participate
3. Patients who speak and read English will be invited to participate.
4. Have the ability to complete the questionnaire.

Exclusion Criteria:

1. Non- English speaking patients.
2. Patients who refuse consent.
3. Patients who are confused or who are cognitively unable to complete the questionnaire.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Szumacher, FRCP(C), Med, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alicikus ZA, Yamada Y, Zhang Z, Pei X, Hunt M, Kollmeier M, Cox B, Zelefsky MJ. Ten-year outcomes of high-dose, intensity-modulated radiotherapy for localized prostate cancer. Cancer. 2011 Apr 1;117(7):1429-37. doi: 10.1002/cncr.25467. Epub 2010 Nov 8. PMID 21425143
- [Background] Michalski JM, Yan Y, Watkins-Bruner D, Bosch WR, Winter K, Galvin JM, Bahary JP, Morton GC, Parliament MB, Sandler HM. Preliminary toxicity analysis of 3-dimensional conformal radiation therapy versus intensity modulated radiation therapy on the high-dose arm of the Radiation Therapy Oncology Group 0126 prostate cancer trial. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):932-8. doi: 10.1016/j.ijrobp.2013.07.041. Epub 2013 Oct 8. PMID 24113055
- [Background] Boersma LJ, van den Brink M, Bruce AM, Shouman T, Gras L, te Velde A, Lebesque JV. Estimation of the incidence of late bladder and rectum complications after high-dose (70-78 GY) conformal radiotherapy for prostate cancer, using dose-volume histograms. Int J Radiat Oncol Biol Phys. 1998 Apr 1;41(1):83-92. doi: 10.1016/s0360-3016(98)00037-6. PMID 9588921
- [Background] Zelefsky MJ, Fuks Z, Happersett L, Lee HJ, Ling CC, Burman CM, Hunt M, Wolfe T, Venkatraman ES, Jackson A, Skwarchuk M, Leibel SA. Clinical experience with intensity modulated radiation therapy (IMRT) in prostate cancer. Radiother Oncol. 2000 Jun;55(3):241-9. doi: 10.1016/s0167-8140(99)00100-0. PMID 10869739
- [Background] Fiorino C, Reni M, Bolognesi A, Cattaneo GM, Calandrino R. Intra- and inter-observer variability in contouring prostate and seminal vesicles: implications for conformal treatment planning. Radiother Oncol. 1998 Jun;47(3):285-92. doi: 10.1016/s0167-8140(98)00021-8. PMID 9681892
- [Background] Fiorino C, Vavassori V, Sanguineti G, Bianchi C, Cattaneo GM, Piazzolla A, Cozzarini C. Rectum contouring variability in patients treated for prostate cancer: impact on rectum dose-volume histograms and normal tissue complication probability. Radiother Oncol. 2002 Jun;63(3):249-55. doi: 10.1016/s0167-8140(01)00469-8. PMID 12142088
- [Background] Fiorino C, Cozzarini C, Vavassori V, Sanguineti G, Bianchi C, Cattaneo GM, Foppiano F, Magli A, Piazzolla A. Relationships between DVHs and late rectal bleeding after radiotherapy for prostate cancer: analysis of a large group of patients pooled from three institutions. Radiother Oncol. 2002 Jul;64(1):1-12. doi: 10.1016/s0167-8140(02)00147-0. PMID 12208568
- [Background] Fiorino C, Gianolini S, Nahum AE. A cylindrical model of the rectum: comparing dose-volume, dose-surface and dose-wall histograms in the radiotherapy of prostate cancer. Phys Med Biol. 2003 Aug 21;48(16):2603-16. doi: 10.1088/0031-9155/48/16/303. PMID 12974577
- [Background] Fokdal L, Honore H, Hoyer M, von der Maase H. Dose-volume histograms associated to long-term colorectal functions in patients receiving pelvic radiotherapy. Radiother Oncol. 2005 Feb;74(2):203-10. doi: 10.1016/j.radonc.2004.11.001. Epub 2004 Nov 25. PMID 15734208
- [Background] Foppiano F, Fiorino C, Frezza G, Greco C, Valdagni R; AIRO National Working Group on Prostate Radiotherapy. The impact of contouring uncertainty on rectal 3D dose-volume data: results of a dummy run in a multicenter trial (AIROPROS01-02). Int J Radiat Oncol Biol Phys. 2003 Oct 1;57(2):573-9. doi: 10.1016/s0360-3016(03)00659-x. PMID 12957271
- [Background] Miralbell R, Taussky D, Rinaldi O, Lomax A, Canales S, Escude L, Nouet P, Ozsoy O, Rouzaud M. Influence of rectal volume changes during radiotherapy for prostate cancer: a predictive model for mild-to-moderate late rectal toxicity. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1280-4. doi: 10.1016/s0360-3016(03)00749-1. PMID 14630262
- [Derived] Dawdy K, Bonin K, Russell S, Ryzynski A, Harth T, Townsend C, Liu S, Chu W, Cheung P, Chung H, Morton G, Vesprini D, Loblaw A, Cao X, Szumacher E. Developing and Evaluating Multimedia Patient Education Tools to Better Prepare Prostate-Cancer Patients for Radiotherapy Treatment (Randomized Study). J Cancer Educ. 2018 Jun;33(3):551-556. doi: 10.1007/s13187-016-1091-5. PMID 27526692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at their initial appointment date or via telephone by our trained research assistant (RA). The RA presented the study rationale to the patients and those who consented were randomly assigned to either the multimedia group or the pamphlet group.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whom Had Proper Preparation After Education Intervention
Description: patients will receive a questionnaire to assess their satisfaction of their appointment. CT scans will be assessed for compliance of preparation based on departmental guidelines and rescans required.
Time Frame: 1 month (patients will be followed until their treatment is complete)
Measure: Number; unit: participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 29 | 29
participants
  Number of patients prepared after intervention | 22 | 22
  Number of patients not prepared after education | 7 | 7

ADVERSE EVENTS:
Time Frame: There were no adverse events to report. This was an education study.
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes